CLINICAL TRIAL: NCT02914639
Title: A Phase I/II Randomized, Double-Masked, Multicenter Clinical Trial Designed to Evaluate the Safety and Exploratory Efficacy of SF0166 Topical Ophthalmic Solution in the Treatment of Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Safety and Exploratory Efficacy Study of SF0166 in the Treatment of Neovascular Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OcuTerra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SF0166-C-002
Record Dates: First submitted 2016-09-01; First posted 2016-09-26 (Estimated); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SF0166 low dose BID (Experimental): SF0166 low dose instilled in study eye BID for 28 days of treatment.
  Interventions: Drug: SF0166 Topical Ophthalmic Solution
- SF0166 high dose BID (Experimental): SF0166 high dose instilled in study eye BID for 28 days of treatment.
  Interventions: Drug: SF0166 Topical Ophthalmic Solution

INTERVENTIONS:
Drug: SF0166 Topical Ophthalmic Solution
  Other Names: OTT166

SUMMARY:
The primary purpose of this study was to evaluate the safety and exploratory efficacy of SF0166 Topical Ophthalmic Solution in patients with Neovascular (wet) Age-related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
This was a prospective, randomized, double-masked, multicenter, Phase I/II clinical study in which 44 eligible subjects with Neovascular Age-related Macular Degeneration (AMD) were randomized to 1 of 2 treatment arms in a 1:1 ratio as follows: SF0166 low dose twice daily (BID) or SF0166 high dose BID.

Study subjects administered the randomly assigned treatment for 28 days. There was an additional 28-day post-treatment follow-up period. Study subjects returned for examination every 2 weeks for 8 weeks (2 months).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 50 years of age or older.
2. Active subfoveal choroidal neovascularization due to Age-related Macular Degeneration (AMD) in the study eye that meet the following criteria:

   * Total lesion ≤12 Macular Photocoagulation Study (MPS) disc areas
   * Choroidal neovascularization (CNV) >50% of lesion area
   * Intraretinal or subretinal fluid due to choroidal neovascularization (CNV) visible on optical coherence tomography (OCT)
   * No atrophy or fibrosis involving the center of the fovea
3. Best-corrected Visual Acuity (BCVA) between 78 and 25 letters, inclusive, in the study eye at the screening/randomization visit using Early Treatment Diabetic Retinopathy Study (ETDRS) testing, with BCVA decrement primarily attributable to neovascular Age-related Macular Degeneration (AMD).
4. Treatment naïve (i.e., no previous anti--vascular endothelial growth factor [VEGF] treatment in the study eye) or previously treated study eye with adequate washout defined below:

   1. Lucentis (ranibizumab): 30-day washout
   2. Avastin (bevacizumab): 30-day washout
   3. Eylea (aflibercept): 60-day washout
   4. Macugen (pegaptanib): 45-day washout
5. Willing and able to return for all study visits.
6. Able to adhere to the study dosing requirements.
7. Understands and signs the written informed consent form.

Exclusion Criteria:

1. Non-study eye best corrected visual acuity (BCVA) worse than 20 letters at the screening/randomization visit using Early Treatment Diabetic Retinopathy Study (ETDRS) testing.
2. Choroidal neovascularization (CNV) in the study eye secondary to other causes (e.g., pathologic myopia, ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, posterior uveitis, or multifocal choroiditis).
3. Previous macular laser photocoagulation or ocular photodynamic therapy in the study eye.
4. Media opacities or abnormalities in the study eye that would preclude visualization of the retina.
5. Other retinal pathologies in the study eye that would interfere with vision.
6. Retinal pigment epithelial (RPE) tear in the study eye.
7. Significant epiretinal membrane, posterior hyaloidal traction, and/or vitreomacular traction in the study eye as determined by optical coherence tomography (OCT) results.
8. Uncontrolled glaucoma or ocular hypertension in the study eye defined as an Intraocular Pressure (IOP) >25 millimeter of mercury (mmHg) regardless of concomitant treatment with IOP lowering medications.
9. Uncontrolled hypertension defined as systolic >180 mmHg or >160 mmHg on 2 consecutive measurements (during the same visit) or diastolic >100 mmHg on optimal medical regimen
10. Previous pars plana vitrectomy in the study eye.
11. Any intraocular surgery in the study eye within 90 days (3 months) prior to study enrollment.
12. Yttrium aluminium garnet (YAG) laser treatment in the study eye within 30 days (1 month) prior to study enrollment.
13. Intravitreal/periocular/topical ocular steroids of any type in the study eye within 90 days (3 months) prior to study enrollment.
14. Concomitant use any topical ophthalmic medications in the study eye, including dry eye or glaucoma medications, unless on a stable dose for at least 90 days (3 months) prior to study enrollment and expected to stay on stable dose throughout study participation. Artificial tears are allowed.
15. Chronic or recurrent uveitis in the study eye.
16. Ongoing ocular infection or inflammation in either eye.
17. A history of cataract surgery complicated by vitreous loss in the study eye.
18. Congenital eye malformations in the study eye.
19. A history of penetrating ocular trauma in the study eye.
20. Mentally handicapped.
21. Females of childbearing potential (i.e., who are not postmenopausal for at least 1 year or surgically sterile for at least 6 weeks prior to Visit 1 - Screening/Randomization) who are lactating, or who are pregnant as determined by a positive urine pregnancy test (UPT) at Visit 1 - Screening/Randomization. Women of childbearing potential must agree to use acceptable methods of birth control throughout the study. Acceptable methods of birth control include tubal ligation, transdermal patch, intrauterine devices/systems, oral/implantable/injectable or contraceptives, sexual abstinence, double barrier method, or vasectomized partner.
22. Participation in any other investigational device or drug clinical research study within 30 days of Visit 1 - Screening/Randomization.
23. Contraindication to the study medications or fluorescein dye.
24. Other ocular pathologies that in the Investigator's opinion would interfere with vision in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foulks, MD, Study Chair — Medical Monitor
Locations (12):
- United States (12):
  - Retinal Research Institute LLC, Phoenix, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates Medical Group, Inc, Mountain View, California
  - Retina Macula Specialists of Miami, LLC, Miami, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - John Kenyon Eye Institute, New Albany, Indiana
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - West Texas Retina Consultants, Abilene, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Spokane Eye Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- SF0166 Low Dose 2.5% BID: SF0166 low dose 2.5% instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
- SF0166 High Dose 5.0% BID: SF0166 high dose 5.0% instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
Period: Overall Study
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Started | 23 | 21
Completed | 23 | 19
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.1 (8.3) | 77.3 (6.1) | 77.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 16 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 20 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Iris Color [Count of Participants; unit: Participants]
  Blue | 10 | 10 | 20
  Brown | 9 | 9 | 18
  Green | 2 | 0 | 2
  Hazel | 2 | 0 | 2
  Gray | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With No Cells Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with no red blood cell counts in the anterior chamber
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: The analysis population includes all randomized participants, 23 in the low dose 2.5% group and 21 in the high dose 5.0% group. One participant in the high dose 5.0% group discontinued prior to Week 2 and one participant in the high dose group discontinued prior to Week 6.
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye) - No Cells Seen | 23 | 21
  Baseline (Fellow Eye) - No Cells Seen | 23 | 21
  Week 2 (Study Eye) - No Cells Seen: number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye) - No Cells Seen | 23 | 20
  Week 2 (Fellow Eye) - No Cells Seen: number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye) - No Cells Seen | 23 | 20
  Week 4 (Study Eye) - No Cells Seen: number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye) - No Cells Seen | 23 | 20
  Week 4 (Fellow Eye) - No Cells Seen: number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye) - No Cells Seen | 23 | 20
  Week 6 (Study Eye) - No Cells Seen: number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye) - No Cells Seen | 23 | 19
  Week 6 (Fellow Eye) - No Cells Seen: number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye) - No Cells Seen | 23 | 19
  Week 8 (Study Eye) - No Cells Seen: number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye) - No Cells Seen | 23 | 19
  Week 8 (Fellow Eye) - No Cells Seen: number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye) - No Cells Seen | 23 | 19

2. Primary Outcome: Number of Subjects With Flare Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with flare in the anterior chamber graded on a scale from 0 (none) to 4 (severe)
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Mild | 1 | 0
  Baseline (Study Eye): None | 22 | 21
  Baseline (Fellow Eye): Mild | 1 | 0
  Baseline (Fellow Eye): None | 22 | 21
  Week 2 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye): Mild | 0 | 0
  Week 2 (Study Eye): None | 23 | 20
  Week 2 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye): Mild | 0 | 0
  Week 2 (Fellow Eye): None | 23 | 20
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): Mild | 1 | 0
  Week 4 (Study Eye): None | 22 | 20
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): Mild | 1 | 0
  Week 4 (Fellow Eye): None | 22 | 20
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): Mild | 0 | 0
  Week 6 (Study Eye): None | 23 | 19
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): Mild | 1 | 0
  Week 6 (Fellow Eye): None | 22 | 19
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): Mild | 0 | 0
  Week 8 (Study Eye): None | 23 | 19
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): Mild | 0 | 0
  Week 8 (Fellow Eye): None | 23 | 19

3. Primary Outcome: Number of Subjects With Absence of Hyphema Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with absence of hyphema
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye) - Absent | 23 | 21
  Baseline (Fellow Eye) - Absent | 23 | 21
  Week 2 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye) - Absent | 23 | 20
  Week 2 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye) - Absent | 23 | 20
  Week 4 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye) - Absent | 23 | 20
  Week 4 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye) - Absent | 23 | 20
  Week 6 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye) - Absent | 23 | 19
  Week 6 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye) - Absent | 23 | 19
  Week 8 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye) - Absent | 23 | 19
  Week 8 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye) - Absent | 23 | 19

4. Primary Outcome: Number of Subjects With Absence of Bulbar Conjunctival Injection Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with absence of bulbar conjunctival injection
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye) - Absent | 23 | 21
  Baseline (Fellow Eye) - Absent | 23 | 21
  Week 2 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye) - Absent | 23 | 20
  Week 2 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye) - Absent | 23 | 20
  Week 4 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye) - Absent | 23 | 20
  Week 4 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye) - Absent | 23 | 20
  Week 6 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye) - Absent | 23 | 19
  Week 6 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye) - Absent | 23 | 19
  Week 8 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye) - Absent | 23 | 19
  Week 8 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye) - Absent | 23 | 19

5. Primary Outcome: Number of Subjects With Absence of Erythema Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with absence of erythema
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye) - Absent | 23 | 21
  Baseline (Fellow Eye) - Absent | 23 | 21
  Week 2 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye) - Absent | 23 | 20
  Week 2 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye) - Absent | 23 | 20
  Week 4 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye) - Absent | 23 | 20
  Week 4 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye) - Absent | 23 | 20
  Week 6 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye) - Absent | 23 | 19
  Week 6 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye) - Absent | 23 | 19
  Week 8 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye) - Absent | 23 | 19
  Week 8 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye) - Absent | 23 | 19

6. Primary Outcome: Number of Subjects With Absence of Edema Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with absence of edema
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye) - Absent | 23 | 21
  Baseline (Fellow Eye) - Absent | 23 | 21
  Week 2 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye) - Absent | 23 | 20
  Week 2 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye) - Absent | 23 | 20
  Week 4 (Study Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye) - Absent | 23 | 20
  Week 4 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye) - Absent | 23 | 19
  Week 6 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye) - Absent | 23 | 19
  Week 6 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye) - Absent | 23 | 19
  Week 8 (Study Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye) - Absent | 23 | 19
  Week 8 (Fellow Eye) - Absent: number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye) - Absent | 23 | 19

7. Primary Outcome: Number of Subjects With Any Lens Opacity Observed Following Slit Lamp Examination From Baseline to Week 8
Description: Number and percentage of subjects with any lens opacity
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Any opacity in the lens | 12 | 7
  Baseline (Study Eye): No opacity in the lens | 11 | 14
  Baseline (Fellow Eye): Any opacity in the lens | 11 | 8
  Baseline (Fellow Eye): No opacity in the lens | 12 | 13
  Week 2 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye): Any opacity in the lens | 12 | 7
  Week 2 (Study Eye): No opacity in the lens | 11 | 13
  Week 2 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye): Any opacity in the lens | 11 | 8
  Week 2 (Fellow Eye): No opacity in the lens | 12 | 12
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): Any opacity in the lens | 12 | 7
  Week 4 (Study Eye): No opacity in the lens | 11 | 13
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): Any opacity in the lens | 11 | 8
  Week 4 (Fellow Eye): No opacity in the lens | 12 | 12
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): Any opacity in the lens | 13 | 8
  Week 6 (Study Eye): No opacity in the lens | 10 | 11
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): Any opacity in the lens | 12 | 9
  Week 6 (Fellow Eye): No opacity in the lens | 11 | 10
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): Any opacity in the lens | 13 | 7
  Week 8 (Study Eye): No opacity in the lens | 10 | 12
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): Any opacity in the lens | 12 | 8
  Week 8 (Fellow Eye): No opacity in the lens | 11 | 11

8. Primary Outcome: Number of Subjects With Abnormal Findings in Optic Nerve Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the optic nerve
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- SF0166High Dose 5.0% BID: SF0166 high dose 5.0% instilled in study eye BID for 28 days of treatment.
  SF0166 Topical Ophthalmic Solution
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Normal | 23 | 19
  Baseline (Study Eye): Abnormal | 0 | 2
  Baseline (Fellow Eye): Normal | 21 | 20
  Baseline (Fellow Eye): Abnormal | 2 | 1
  Week 2 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye): Normal | 23 | 19
  Week 2 (Study Eye): Abnormal | 0 | 1
  Week 2 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye): Normal | 21 | 19
  Week 2 (Fellow Eye): Abnormal | 2 | 1
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): Normal | 23 | 19
  Week 4 (Study Eye): Abnormal | 0 | 1
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): Normal | 21 | 19
  Week 4 (Fellow Eye): Abnormal | 2 | 1
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): Normal | 23 | 18
  Week 6 (Study Eye): Abnormal | 0 | 1
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): Normal | 21 | 18
  Week 6 (Fellow Eye): Abnormal | 2 | 1
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): Normal | 23 | 18
  Week 8 (Study Eye): Abnormal | 0 | 1
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): Normal | 21 | 18
  Week 8 (Fellow Eye): Abnormal | 2 | 1

9. Primary Outcome: Number of Subjects With Abnormal Findings in Vitreous Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the vitreous
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Normal | 16 | 8
  Baseline (Study Eye): Abnormal | 7 | 13
  Baseline (Fellow Eye): Normal | 15 | 6
  Baseline (Fellow Eye): Abnormal | 8 | 15
  Week 2 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye): Normal | 15 | 7
  Week 2 (Study Eye): Abnormal | 8 | 13
  Week 2 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye): Normal | 15 | 6
  Week 2 (Fellow Eye): Abnormal | 8 | 14
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): Normal | 15 | 7
  Week 4 (Study Eye): Abnormal | 8 | 13
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): Normal | 15 | 6
  Week 4 (Fellow Eye): Abnormal | 8 | 14
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): Normal | 15 | 7
  Week 6 (Study Eye): Abnormal | 8 | 12
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): Normal | 15 | 6
  Week 6 (Fellow Eye): Abnormal | 8 | 13
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): Normal | 15 | 8
  Week 8 (Study Eye): Abnormal | 8 | 11
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): Normal | 15 | 7
  Week 8 (Fellow Eye): Abnormal | 8 | 12

10. Primary Outcome: Number of Subjects With Abnormal Findings in Fundus Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the fundus
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Normal | 19 | 18
  Baseline (Study Eye): Abnormal | 4 | 3
  Baseline (Fellow Eye): Normal | 19 | 18
  Baseline (Fellow Eye): Abnormal | 4 | 3
  Week 2 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye): Normal | 19 | 16
  Week 2 (Study Eye): Abnormal | 4 | 4
  Week 2 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye): Normal | 19 | 17
  Week 2 (Fellow Eye): Abnormal | 4 | 3
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): Normal | 19 | 17
  Week 4 (Study Eye): Abnormal | 4 | 3
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): Normal | 19 | 17
  Week 4 (Fellow Eye): Abnormal | 4 | 3
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): Normal | 19 | 16
  Week 6 (Study Eye): Abnormal | 4 | 3
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): Normal | 19 | 16
  Week 6 (Fellow Eye): Abnormal | 4 | 3
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): Normal | 19 | 16
  Week 8 (Study Eye): Abnormal | 4 | 3
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): Normal | 19 | 16
  Week 8 (Fellow Eye): Abnormal | 4 | 3

11. Primary Outcome: Number of Subjects With Abnormal Findings in Macula/Choroid Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the macula/choroid
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Normal | 23 | 21
  Baseline (Study Eye): Abnormal | 0 | 0
  Baseline (Fellow Eye): Normal | 0 | 1
  Baseline (Fellow Eye): Abnormal | 23 | 20
  Week 2 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye): Normal | 0 | 0
  Week 2 (Study Eye): Abnormal | 23 | 20
  Week 2 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye): Normal | 1 | 1
  Week 2 (Fellow Eye): Abnormal | 22 | 19
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): Normal | 23 | 20
  Week 4 (Study Eye): Abnormal | 0 | 0
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): Normal | 1 | 0
  Week 4 (Fellow Eye): Abnormal | 22 | 20
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): Normal | 0 | 0
  Week 6 (Study Eye): Abnormal | 23 | 19
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): Normal | 1 | 0
  Week 6 (Fellow Eye): Abnormal | 22 | 19
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): Normal | 23 | 19
  Week 8 (Study Eye): Abnormal | 0 | 0
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): Normal | 1 | 0
  Week 8 (Fellow Eye): Abnormal | 22 | 19

12. Primary Outcome: Number of Subjects With Abnormal Findings in Vessels Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with abnormal findings in the retinal vessels
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Normal | 20 | 18
  Baseline (Study Eye): Abnormal | 3 | 3
  Baseline (Fellow Eye): Normal | 22 | 18
  Baseline (Fellow Eye): Abnormal | 1 | 3
  Week 2 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Study Eye): Normal | 20 | 17
  Week 2 (Study Eye): Abnormal | 3 | 3
  Week 2 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 2 (Fellow Eye): Normal | 22 | 17
  Week 2 (Fellow Eye): Abnormal | 1 | 3
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): Normal | 19 | 17
  Week 4 (Study Eye): Abnormal | 4 | 3
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): Normal | 22 | 17
  Week 4 (Fellow Eye): Abnormal | 1 | 3
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): Normal | 20 | 16
  Week 6 (Study Eye): Abnormal | 3 | 3
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): Normal | 22 | 16
  Week 6 (Fellow Eye): Abnormal | 1 | 3
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): Normal | 19 | 16
  Week 8 (Study Eye): Abnormal | 4 | 3
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): Normal | 22 | 16
  Week 8 (Fellow Eye): Abnormal | 1 | 3

13. Primary Outcome: Cup:Disc Ratio of Subjects Following Fundus Examination From Baseline to Week 8
Description: Number and percentage of subjects with specified Cup:Disc ratio in the range from 0.1 to 0.9 with the higher number being worse
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: The analysis population includes all randomized participants, 23 in the low dose 2.5% group and 21 in the high dose 5.0% group. One participant in the low dose group 2.5% group did not have values recorded at Baseline or Week 2 for either the study eye or the fellow eye. One participant in the high dose 5.0% group discontinued prior to Week 2 and one participant in the high dose group discontinued prior to Week 6.
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): number analyzed (Participants) | 22 | 21
  Baseline (Study Eye): 0.10 | 1 | 2
  Baseline (Study Eye): 0.20 | 8 | 8
  Baseline (Study Eye): 0.30 | 8 | 8
  Baseline (Study Eye): 0.40 | 2 | 2
  Baseline (Study Eye): 0.50 | 1 | 0
  Baseline (Study Eye): 0.70 | 0 | 0
  Baseline (Study Eye): 0.75 | 0 | 1
  Baseline (Study Eye): 0.85 | 1 | 0
  Baseline (Study Eye): 0.90 | 1 | 0
  Baseline (Fellow Eye): number analyzed (Participants) | 22 | 21
  Baseline (Fellow Eye): 0.10 | 1 | 3
  Baseline (Fellow Eye): 0.20 | 7 | 6
  Baseline (Fellow Eye): 0.30 | 8 | 7
  Baseline (Fellow Eye): 0.40 | 1 | 4
  Baseline (Fellow Eye): 0.50 | 3 | 1
  Baseline (Fellow Eye): 0.70 | 0 | 0
  Baseline (Fellow Eye): 0.75 | 1 | 0
  Baseline (Fellow Eye): 0.85 | 0 | 0
  Baseline (Fellow Eye): 0.90 | 1 | 0
  Week 2 (Study Eye): number analyzed (Participants) | 22 | 20
  Week 2 (Study Eye): 0.10 | 1 | 2
  Week 2 (Study Eye): 0.20 | 8 | 8
  Week 2 (Study Eye): 0.30 | 8 | 7
  Week 2 (Study Eye): 0.40 | 2 | 2
  Week 2 (Study Eye): 0.50 | 1 | 0
  Week 2 (Study Eye): 0.70 | 0 | 0
  Week 2 (Study Eye): 0.75 | 0 | 1
  Week 2 (Study Eye): 0.85 | 1 | 0
  Week 2 (Study Eye): 0.90 | 1 | 0
  Week 2 (Fellow Eye): number analyzed (Participants) | 22 | 20
  Week 2 (Fellow Eye): 0.10 | 1 | 3
  Week 2 (Fellow Eye): 0.20 | 7 | 6
  Week 2 (Fellow Eye): 0.30 | 8 | 6
  Week 2 (Fellow Eye): 0.40 | 1 | 4
  Week 2 (Fellow Eye): 0.50 | 3 | 1
  Week 2 (Fellow Eye): 0.70 | 1 | 0
  Week 2 (Fellow Eye): 0.75 | 0 | 0
  Week 2 (Fellow Eye): 0.85 | 0 | 0
  Week 2 (Fellow Eye): 0.90 | 1 | 0
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Study Eye): 0.10 | 1 | 2
  Week 4 (Study Eye): 0.20 | 8 | 8
  Week 4 (Study Eye): 0.30 | 9 | 7
  Week 4 (Study Eye): 0.40 | 2 | 2
  Week 4 (Study Eye): 0.50 | 1 | 0
  Week 4 (Study Eye): 0.70 | 0 | 0
  Week 4 (Study Eye): 0.75 | 0 | 1
  Week 4 (Study Eye): 0.85 | 1 | 0
  Week 4 (Study Eye): 0.90 | 1 | 0
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 20
  Week 4 (Fellow Eye): 0.10 | 1 | 3
  Week 4 (Fellow Eye): 0.20 | 7 | 6
  Week 4 (Fellow Eye): 0.30 | 9 | 6
  Week 4 (Fellow Eye): 0.40 | 1 | 4
  Week 4 (Fellow Eye): 0.50 | 3 | 1
  Week 4 (Fellow Eye): 0.70 | 0 | 0
  Week 4 (Fellow Eye): 0.75 | 1 | 0
  Week 4 (Fellow Eye): 0.85 | 0 | 0
  Week 4 (Fellow Eye): 0.90 | 1 | 0
  Week 6 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Study Eye): 0.10 | 1 | 2
  Week 6 (Study Eye): 0.20 | 8 | 9
  Week 6 (Study Eye): 0.30 | 9 | 6
  Week 6 (Study Eye): 0.40 | 2 | 1
  Week 6 (Study Eye): 0.50 | 1 | 0
  Week 6 (Study Eye): 0.70 | 0 | 0
  Week 6 (Study Eye): 0.75 | 0 | 1
  Week 6 (Study Eye): 0.85 | 1 | 0
  Week 6 (Study Eye): 0.90 | 1 | 0
  Week 6 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 6 (Fellow Eye): 0.10 | 1 | 3
  Week 6 (Fellow Eye): 0.20 | 7 | 7
  Week 6 (Fellow Eye): 0.30 | 9 | 5
  Week 6 (Fellow Eye): 0.40 | 1 | 3
  Week 6 (Fellow Eye): 0.50 | 3 | 1
  Week 6 (Fellow Eye): 0.70 | 0 | 0
  Week 6 (Fellow Eye): 0.75 | 1 | 0
  Week 6 (Fellow Eye): 0.85 | 0 | 0
  Week 6 (Fellow Eye): 0.90 | 1 | 0
  Week 8 (Study Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Study Eye): 0.10 | 1 | 2
  Week 8 (Study Eye): 0.20 | 8 | 9
  Week 8 (Study Eye): 0.30 | 9 | 6
  Week 8 (Study Eye): 0.40 | 2 | 1
  Week 8 (Study Eye): 0.50 | 1 | 0
  Week 8 (Study Eye): 0.70 | 0 | 0
  Week 8 (Study Eye): 0.75 | 0 | 1
  Week 8 (Study Eye): 0.85 | 1 | 0
  Week 8 (Study Eye): 0.90 | 1 | 0
  Week 8 (Fellow Eye): number analyzed (Participants) | 23 | 19
  Week 8 (Fellow Eye): 0.10 | 1 | 2
  Week 8 (Fellow Eye): 0.20 | 7 | 8
  Week 8 (Fellow Eye): 0.30 | 9 | 5
  Week 8 (Fellow Eye): 0.40 | 1 | 3
  Week 8 (Fellow Eye): 0.50 | 3 | 1
  Week 8 (Fellow Eye): 0.70 | 0 | 0
  Week 8 (Fellow Eye): 0.75 | 1 | 0
  Week 8 (Fellow Eye): 0.85 | 0 | 0
  Week 8 (Fellow Eye): 0.90 | 1 | 0

14. Primary Outcome: Number of Subjects With Abnormal Findings Following A Fluorescein Angiogram at Week 4 Compared to Baseline
Description: Number and percentage of subjects with abnormal fluorescein angiogram findings
Time Frame: Baseline and Week 4
Population: The analysis population includes all randomized participants, 23 in the low dose 2.5% group and 21 in the high dose 5.0% group. One participant in the high dose 5.0% group discontinued prior to Week 4. Angiograms were not obtained for two participants in the high dose 5.0% group at Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
Participants
  Baseline (Study Eye): Abnormal | 23 | 21
  Baseline (Study Eye): Normal | 0 | 0
  Baseline (Fellow Eye): Abnormal | 23 | 18
  Baseline (Fellow Eye): Normal | 0 | 3
  Week 4 (Study Eye): number analyzed (Participants) | 23 | 18
  Week 4 (Study Eye): Abnormal | 23 | 18
  Week 4 (Study Eye): Normal | 0 | 0
  Week 4 (Fellow Eye): number analyzed (Participants) | 23 | 18
  Week 4 (Fellow Eye): Abnormal | 20 | 15
  Week 4 (Fellow Eye): Normal | 3 | 3

15. Primary Outcome: Change in Intraocular Pressure From Baseline to Week 8
Description: Mean and standard deviation of change from Baseline in intra-ocular pressure
Time Frame: Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 23 | 21
mmHg
  Change from Baseline in Study Eye at Week 2: number analyzed (Participants) | 23 | 20
  Change from Baseline in Study Eye at Week 2 | 0.1 (3.2) | 0.5 (2.8)
  Change from Baseline in Non-Study Eye at Week 2: number analyzed (Participants) | 23 | 20
  Change from Baseline in Non-Study Eye at Week 2 | 0.3 (3.1) | 1.4 (2.6)
  Change from Baseline in Study Eye at Week 4: number analyzed (Participants) | 23 | 20
  Change from Baseline in Study Eye at Week 4 | -1.0 (3.0) | 0.5 (3.5)
  Change from Baseline in Non-Study Eye at Week 4: number analyzed (Participants) | 23 | 20
  Change from Baseline in Non-Study Eye at Week 4 | -0.7 (4.1) | 0.7 (2.6)
  Change from Baseline in Study Eye at Week 6: number analyzed (Participants) | 23 | 19
  Change from Baseline in Study Eye at Week 6 | -0.4 (3.2) | 0.9 (3.4)
  Change from Baseline in Non-Study Eye at Week 6: number analyzed (Participants) | 23 | 19
  Change from Baseline in Non-Study Eye at Week 6 | -0.7 (3.3) | 0.2 (3.1)
  Change from Baseline in Study Eye at Week 8: number analyzed (Participants) | 23 | 19
  Change from Baseline in Study Eye at Week 8 | -0.5 (4.0) | 0.4 (3.3)
  Change from Baseline in Non-Study Eye at Week 8: number analyzed (Participants) | 23 | 19
  Change from Baseline in Non-Study Eye at Week 8 | 0.3 (3.7) | 0.6 (3.0)

16. Primary Outcome: Change in Study Eye Central Retinal Thickness (CRT) From Baseline (Day 0) to Week 8
Description: Results are mean plus standard deviation
Time Frame: Week 2, Week 4, Week 6 and Week 8
Population: The analysis population is the per protocol population with 22 participants in the low dose 2.5% and 19 participants in the high dose 5.0% group at Baseline. Prior to Week 6, two participants in the low dose 2.5% group and three in the high dose 5.0% group were given rescue medication; the data excluded for Week 6 and Week 8. Three participants in the high dose 5.0% group were rescued prior to Week 8; the data for Week 8 are excluded.
Measure: Mean (Standard Deviation); unit: change from baseline
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 19
change from baseline
  Change from Baseline at Week 2 | -1.6 (36.2) | 3.8 (25.4)
  Change from Baseline at Week 4 | -1.3 (83.0) | 13.8 (54.0)
  Change from Baseline at Week 6: number analyzed (Participants) | 20 | 16
  Change from Baseline at Week 6 | 26.1 (117.0) | -8.2 (32.8)
  Change from Baseline at Week 8: number analyzed (Participants) | 20 | 13
  Change from Baseline at Week 8 | 27.5 (105.1) | -6.9 (35.9)

17. Secondary Outcome: Change in Best-corrected Visual Acuity (BCVA) From Baseline (Day 0) at Week 4 and Week 8
Description: Results are mean plus standard deviation in per protocol population.
Time Frame: Week 2, Week 4, Week 6, and Week 8
Population: IThe analysis population is the per protocol population with 22 participants in the low dose 2.5% and 19 participants in the high dose 5.0% group at Baseline. Prior to Week 6, two participants in the low dose 2.5% group and three in the high dose 5.0% group were given rescue medication; the data excluded for Week 6 and Week 8. Three participants in the high dose 5.0% group were rescued prior to Week 8; the data for Week 8 are excluded.
Measure: Mean (Standard Deviation); unit: change from baseline
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
Number analyzed (Participants) | 22 | 19
change from baseline
  Change from Baseline at Week 2 | 2.8 (7.1) | 2.8 (5.0)
  Change from Baseline at Week 4 | 2.5 (6.7) | 1.7 (6.5)
  Change from Baseline at Week 6: number analyzed (Participants) | 20 | 16
  Change from Baseline at Week 6 | 1.3 (4.3) | 2.4 (9.0)
  Change from Baseline at Week 8: number analyzed (Participants) | 20 | 13
  Change from Baseline at Week 8 | 1.0 (5.4) | 1.9 (9.4)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | SF0166 Low Dose 2.5% BID | SF0166 High Dose 5.0% BID
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/21
Other Adverse Events (participants affected / at risk) | 2/23 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SF0166 Low Dose 2.5% BID (N=23) | SF0166 High Dose 5.0% BID (N=21)
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SF0166 Low Dose 2.5% BID (N=23) | SF0166 High Dose 5.0% BID (N=21)
Heart valve incompetence (Cardiac disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02914639/Prot_SAP_000.pdf